CLINICAL TRIAL: NCT04115319
Title: A Randomized, Double-blind, Active Comparator-Controlled Study to Evaluate the Long-term Safety and Tolerability of SEP-363856 in Subjects With Schizophrenia
Brief Title: A Study of the Long-term Safety and Tolerability of an Investigational Drug in People With Schizophrenia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP361-304; 2019-002259-40 (EudraCT Number)
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2024-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-blind, Active Comparator-Controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SEP363856 (Experimental): SEP363856 50mg, 75mg, 100mg, flexibly dosed once daily capsule
  Interventions: Drug: SEP363856
- quetiapine XR (Active Comparator): quetiapine XR, 400, 600, 800 mg, flexibly dosed once daily capsule
  Interventions: Drug: quetiapine XR

INTERVENTIONS:
Drug: SEP363856 — SEP-363856, 50mg, 75mg, 100mg, flexibly dosed once daily capsule
  Arms: SEP363856
Drug: quetiapine XR — quetiapine XR, 400, 600, 800 mg, flexibly dosed once daily capsule
  Other Names: Seroquel XR
  Arms: quetiapine XR

SUMMARY:
A clinical study to evaluate the long-term safety and tolerability of an investigational drug in people with schizophrenia.

This study is accepting male and female participants between 18 years old -65 years old who have been diagnosed with schizophrenia. This study will be conducted in approximately 50 study centers worldwide. The study will last approximately 57 weeks.

DETAILED DESCRIPTION:
This is a 52-week, multicenter, randomized, double-blind, parallel-group, flexible-dose study designed to evaluate the long-term safety and tolerability of SEP-363856 (50 to 100 mg/day) compared with quetiapine XR (400 to 800 mg/day) in clinically stable adult participants with schizophrenia. This study is projected to randomize a least 300 participants to two treatment groups (SEP-363856 50 to 100 mg/day or quetiapine XR 400 to 800 mg/day) in a 2:1 ratio. Study drug will be taken once a day and may be taken without food or with a light meal.

Sumitomo Pharma America Inc. was the former Sponsor and conducted this study. Sumitomo was responsible for analysis and clinical study report (CSR) completion. Otsuka took over study after IND was transferred and is concluding activities with registry postings.

ELIGIBILITY:
Inclusion criteria:

The main inclusion criteria include, but are not limited to the following:

* Male or female participant between 18 to 65 years of age (inclusive) at the time of consent.
* Participant meets DSM-5 criteria for a diagnosis of schizophrenia as established by clinical interview at screening (using the DSM-5 as a reference and confirmed using the SCID-CT). The time since the participant's diagnosis must be ≥ 1 year prior to Screening.
* Participant must have a CGI-S score ≤ 4 at Screening and Baseline.
* Participant must have a PANSS total score ≤ 80 at Screening and Baseline.
* Participant is judged to be clinically stable (i.e., no evidence of an acute exacerbation) by the Investigator for at least 8 weeks prior to Screening.
* Participant has had no change in antipsychotic medication(s) (minor dose adjustments for tolerability purposes are permitted) for at least 6 weeks prior to Screening.
* Participants taking an antipsychotic agent at Screening may participate in this study only if there are signs of intolerability or lack of efficacy of the current antipsychotic (as determined by the Investigator).
* Participant is, in the opinion of the Investigator, generally healthy based on Screening medical history, PE, neurological examination, vital signs, electrocardiogram (ECG) and clinical laboratory values (hematology, chemistry and urinalysis).

Exclusion criteria:

Main exclusion criteria include, but are not limited to:

* Participant was hospitalized for a psychiatric illness within the 8 weeks prior to Screening.
* Participant has a current DSM-5 diagnosis or presence of symptoms consistent with a DSM-5 diagnosis other than schizophrenia. Exclusionary disorders include but are not limited to alcohol use disorder (within past 12 months), substance (other than nicotine or caffeine) use disorder within past 12 months, or lifetime history of significant substance abuse that, in the opinion of the Investigator or Sponsor, may have had a significant and potentially permanent impact on the brain or other body systems, major depressive disorder, schizoaffective disorder, ,bipolar I or II disorder, obsessive compulsive disorder, and posttraumatic stress disorder, symptoms of mild to moderate mood dysphoria or anxiety are allowed so long as theses symptoms are not the primary focus of treatment.
* Participant is judged to be resistant to antipsychotic treatment by the Investigator, based on failure to respond to 2 or more marketed antipsychotic agents within a 1-year period prior to Screening, given at adequate dose as per labeling, for at least 4 weeks.
* Participant answers "yes" to "Suicidal Ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at Screening (i.e., in the past one month) or at Baseline (i.e., since last visit).
* Participant is at significant risk of harming self or others based on Investigator's judgment.
* Participant has attempted suicide within 6 months prior to Screening.
* Participant has received treatment with a psychotropic medication or herbal supplement within 3 days or 5 half-lives (whichever is longer)
* Participant has been treated with quetiapine or quetiapine XR within the 6 weeks prior to Screening or has a history of inadequate response or intolerability to quetiapine or quetiapine XR.
* Participant has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the participant's ability to complete and/or participate in the study.
* Participant has any clinically significant abnormal laboratory value(s) at Screening as determined by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (18):
  - Research Site, Cerritos, California
  - Research Site, Oakland, California
  - Research Site, Oceanside, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Lincolnwood, Illinois
  - Research Site, Shreveport, Louisiana
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Cedarhurst, New York
  - Research Site, Jamaica, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, North Canton, Ohio
- Romania (3):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Iași
- Russia (9):
  - Research Site, Arkhangelsk
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Smolensk
  - Research Site, Stavropol
  - Research Site, Tomsk
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Ukraine (6):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Smila
  - Research Site, Ternopil
  - Research Site, Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at investigational sites in Russia, US, Romania and Ukraine from 21 Nov 2019 to 30 Dec 2022.
Pre-assignment Details: A total of 461 participants were screened, of which 305 participants were randomized and 303 participants received either SEP-363856 (N = 201) or quetiapine XR (N = 102).
Groups:
- SEP-363856 50 to 100 mg/Day: Participants received flexible doses of SEP-363856 50 to 100 milligram per day (mg/day), orally, once daily (QD) up to Week 52. The dose was titrated up from 50 mg/day on Days 1 to 3, to 75 mg/day on Days 4 to 7. Beginning Day 8, the dose was adjusted within the range of 50 mg/day to 100 mg/day in 25 mg increments (i.e. 50, 75, or 100 mg/day) up to Week 52.
- Quetiapine XR 400 to 800 mg/Day: Participants received flexible doses of quetiapine XR 300 to 800 mg/day, orally, QD up to Week 52. The dose was titrated up from 300 mg/day on Days 1 to 2, followed by 400 mg/day on Days 3 to 4, to 600 mg/day on Days 5 to 7. Beginning Day 8, the dose was adjusted within the range of 400 mg/day to 800 mg/day in 200 mg increments (i.e. 400, 600, or 800 mg/day) up to Week 52.
Period: Overall Study
Arm/Group | SEP-363856 50 to 100 mg/Day | Quetiapine XR 400 to 800 mg/Day
Started | 203 | 102
Completed | 105 | 57
Not Completed | 98 | 45
Not completed — Randomized, but Withdrawn From Study Prior to Treatment | 2 | 0
Not completed — Withdrawal by participant | 17 | 9
Not completed — Geopolitical Conflict Related | 2 | 1
Not completed — COVID-19 Related | 1 | 0
Not completed — Adverse Event | 48 | 21
Not completed — Noncompliance with Study Drug | 5 | 1
Not completed — Lack of Efficacy | 6 | 2
Not completed — Lost to Follow-up | 6 | 7
Not completed — Protocol Deviation | 5 | 1
Not completed — Participant relocated | 5 | 2
Not completed — Personal Reasons | 0 | 1
Not completed — Deemed Unsuitable for Participation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants that were enrolled and received at least 1 dose of study drug during the 52-week treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | SEP-363856 50 to 100 mg/Day | Quetiapine XR 400 to 800 mg/Day | Total
Number analyzed (Participants) | 201 | 102 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (11.77) | 38.4 (12.66) | 39.7 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 37 | 125
  Male | 113 | 65 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 193 | 98 | 291
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 28 | 75
  White | 150 | 73 | 223
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 2 | 1 | 3
  United States | 74 | 39 | 113
  Ukraine | 42 | 21 | 63
  Russia | 83 | 41 | 124

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Events (AEs) Leading to Study Discontinuation
Description: An AE was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Untoward medical occurrences that occured after first administration of study drug were considered AEs. A SAE is an AE that meets one or more criteria: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, or is a congenital anomaly or birth defect.
Time Frame: From first dose of the study drug up to 7 days after last dose of study drug (Up to 53 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SEP-363856 50 to 100 mg/Day | Quetiapine XR 400 to 800 mg/Day
Number analyzed (Participants) | 201 | 102
Participants
  AEs | 153 | 77
  SAEs | 16 | 0
  AEs Leading to Trial Discontinuation | 48 | 21

ADVERSE EVENTS:
Time Frame: From first dose of the study drug up to 7 days after last dose of study drug (Up to 53 weeks)
Description: Safety population included all participants that were enrolled and received at least 1 dose of the study drug during the 52-week treatment period.
Arm/Group | SEP-363856 50 to 100 mg/Day | Quetiapine XR 400 to 800 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/102
Serious Adverse Events (participants affected / at risk) | 16/201 | 0/102
Other Adverse Events (participants affected / at risk) | 103/201 | 55/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-363856 50 to 100 mg/Day (N=201) | Quetiapine XR 400 to 800 mg/Day (N=102)
Schizophrenia (Psychiatric disorders) | 10 (10) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-363856 50 to 100 mg/Day (N=201) | Quetiapine XR 400 to 800 mg/Day (N=102)
Weight decreased (Investigations) | 11 (11) | 1 (1)
Weight increased (Investigations) | 9 (9) | 11 (11)
Akathisia (Nervous system disorders) | 14 (15) | 2 (2)
Dizziness (Nervous system disorders) | 16 (18) | 5 (5)
Headache (Nervous system disorders) | 20 (29) | 8 (8)
Somnolence (Nervous system disorders) | 12 (13) | 21 (24)
Asthenia (General disorders) | 5 (6) | 9 (10)
Constipation (Gastrointestinal disorders) | 7 (8) | 12 (16)
Nausea (Gastrointestinal disorders) | 13 (13) | 4 (5)
Anxiety (Psychiatric disorders) | 27 (41) | 10 (12)
Insomnia (Psychiatric disorders) | 30 (38) | 11 (13)
Schizophrenia (Psychiatric disorders) | 21 (23) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT04115319/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT04115319/SAP_001.pdf